CLINICAL TRIAL: NCT03304262
Title: Metaplasticity in the Human Motor Cortex: Validation of an Experimental Design and Comparison of Motor Outcome Measure Sensitivity to Change
Brief Title: Metaplasticity Experimental Design and Comparison of Motor Outcome Measure Sensitivity to Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Sarah Pirio Richardson, Assistant Professor of Neurology, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16-410
Record Dates: First submitted 2017-09-21; First posted 2017-10-06 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Metaplasticity; Motor excitability; rTMS; tDCS

STUDY DESIGN:
Intervention Model Description: This is a randomized, sham-controlled, double blinded crossover trial.
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded to treatment group, investigator administering tDCS will be blinded to which treatment arm subject is assigned to, and the data analyst will be conducting analysis off site and is different than investigator applying stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Cathodal tDCS + rTMS then Anodal tDCS + rTMS then Sham tDCS + rTMS (Active Comparator): Participant will receive 10 minutes of cathodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of anodal tDCS and rTMS for 900 1Hz pulses at 0.85 RMT. After 1 week washout, participant will receive 10 minutes of sham tDCS and rTMS for 900 1 Hz pulses at 0.85 RMT.
  Interventions: Device: rTMS
- Anodal tDCS + rTMS then Sham tDCS + rTMS then Cathodal tDCS + rTMS (Active Comparator): Participant will receive 10 minutes of anodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of sham tDCS and rTMS for 900 1 Hz pulses at 0.85 RMT. After 1 week washout, participant will receive 10 minutes of cathodal tDCS and rTMS for 900 1 Hz pulses at 0.85 RMT.
  Interventions: Device: rTMS
- Sham tDCS + rTMS then Cathodal tDCS + rTMS then Anodal tDCS + rTMS (Sham Comparator): Participant will receive 10 minutes of sham tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of cathodal tDCS and rTMS for 900 1 Hz pulses at 0.85 RMT. After 1 week washout, participant will receive 10 minutes of anodal tDCS and rTMS for 900 1 Hz pulses at 0.85 RMT.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
  Other Names: rapid transcranial magnetic stimulation

SUMMARY:
The overall objective is to validate the methodology of a metaplasticity experimental design by assessing change in motor excitability after administration of priming transcranial direct current stimulation (tDCS) followed by repetitive transcranial magnetic stimulation (rTMS) in healthy human participants.

DETAILED DESCRIPTION:
The overall objective is to validate the methodology of a metaplasticity experimental design by assessing change in motor excitability after administration of priming transcranial direct current stimulation (tDCS) followed by repetitive transcranial magnetic stimulation (rTMS) in healthy human participants. Our primary objective is to compare pre- and post-measures of cortical excitability before priming tDCS (anodal, cathodal or sham) [M1], directly after priming tDCS [M2], directly after inhibitory rTMS [M3], and 10 minutes after inhibitory rTMS [M4]. Our secondary objective is to evaluate the sensitivity of motor excitability outcome measures response to the noninvasive neurostimulation (e.g. rTMS and tDCS). We also aim to compare pre- and post- measures of cortical excitability after inhibitory and excitatory priming of the motor cortex, and to evaluate the sensitivity of motor outcome measures to changes in cortical plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age (all genders, races, ethnicity)
* Must have no current psychiatric or neurologic issues
* Must not have any conditions listed in exclusion criteria
* Must be fluent in English

Exclusion Criteria:

* History of major psychiatric illness
* Actively using neuropsychoactive medication
* Legal or mental incompetency
* Substance use disorder, abuse or dependence, with active use within the last three months
* Significant medical or neurological illness
* Prior neurosurgical illness
* Prior neurosurgical procedure
* History of seizure
* History of ECT or TMS treatment within the past there months
* Presence of a pacemaker, implanted medical pump or device, metal plate, or metal object in skull or eye (including shunts, dental implants, facial tattoos with metallic ink)
* Pregnant women

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pirio Richardson, M.D., Principal Investigator — University of New Mexico; Davin Quinn, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover design, in which each participant came in three times and was randomly assigned to each intervention with a wash-out period in between.
Groups:
- Cathodal tDCS + rTMS Then Anodal tDCS + rTMS Then Sham tDCS + rTMS: Participant will receive 10 minutes of cathodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of anodal tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of sham tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
- Anodal tDCS + rTMS Then Sham tDCS + rTMS Then Cathodal tDCS + rTMS: Participant will receive 10 minutes of anodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of sham tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of cathodal tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
- Sham tDCS + rTMS Then Cathodal tDCS + rTMS Then Anodal tDCS + rTMS: Participant will receive 10 minutes of sham tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of cathodal tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2. After 1 week washout, participant will receive 10 minutes of anodal tDCS between M1 and M2 timepoints, and rTMS for 900 1 Hz pulses at 0.85 Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
Period: Overall Study
Arm/Group | Cathodal tDCS + rTMS Then Anodal tDCS + rTMS Then Sham tDCS + rTMS | Anodal tDCS + rTMS Then Sham tDCS + rTMS Then Cathodal tDCS + rTMS | Sham tDCS + rTMS Then Cathodal tDCS + rTMS Then Anodal tDCS + rTMS
Started | 4 | 5 | 4
Completed | 4 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cathodal tDCS + rTMS Then Anodal tDCS + rTMS Then Sham tDCS + rTMS | Anodal tDCS + rTMS Then Sham tDCS + rTMS Then Cathodal tDCS + rTMS | Sham tDCS + rTMS Then Cathodal tDCS + rTMS Then Anodal tDCS + rTMS | Total
Number analyzed (Participants) | 4 | 5 | 4 | 13
Age, Continuous [Mean (Full Range); unit: years] | 35.54 [23 to 52] | 35.54 [28 to 46] | 35.54 [25 to 36] | 35.54 [23 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 8
  Not Hispanic or Latino | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 4 | 2 | 9
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in MEP Amplitude
Description: Percent Change in MEP amplitude over the first dorsal interosseous (FDI) muscle of the right hand
Time Frame: assessed and reported throughout study completion pre- and post- intervention approximately 30 minutes
Measure: Mean (Full Range); unit: Percent Change
Groups:
- Cathodal tDCS + rTMS: Participant will receive 10 minutes of cathodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
- Anodal tDCS + rTMS: Participant will receive 10 minutes of anodal tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
- Sham tDCS + rTMS: Participant will receive 10 minutes of sham tDCS between M1 and M2 timepoints, and rTMS for 900 1Hz pulses at 0.85 of Resting Motor Threshold at M2.
  rTMS: Between time point M2 and M3, participant will receive 900 pulses of rTMS at 1Hz at 0.85 of M2 resting motor threshold.
Arm/Group | Cathodal tDCS + rTMS | Anodal tDCS + rTMS | Sham tDCS + rTMS
Number analyzed (Participants) | 13 | 13 | 13
Percent Change | 1.19 [0.43 to 5.65] | 1.06 [0.33 to 2.03] | 1.38 [0.19 to 2.82]

2. Secondary Outcome: Cortical Silent Period
Description: Change in length of CSP
Time Frame: tDCS + rTMS assessed and reported pre and post (approximately 10 minutes)
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Cathodal tDCS + rTMS | Anodal tDCS + rTMS | Sham tDCS + rTMS
Number analyzed (Participants) | 13 | 13 | 13
Percent change | 1.02 [0.88 to 1.23] | 1.01 [0.88 to 1.13] | 0.99 [.88 to 1.08]

3. Secondary Outcome: Simple Reaction Time
Description: Participants will perform a simple reaction time task. This will be measured in seconds of response after a stimulus. The final outcome will be percent change in the reaction time from pre- to post- intervention.
Time Frame: The final outcome will be percent change in the reaction time from pre- to post- intervention.
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Cathodal tDCS + rTMS | Anodal tDCS + rTMS | Sham tDCS + rTMS
Number analyzed (Participants) | 13 | 13 | 13
Percent change | 1.01 [0.94 to 1.15] | 1.02 [0.91 to 1.19] | 1.02 [0.9 to 1.16]

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Cathodal tDCS + rTMS | Anodal tDCS + rTMS | Sham tDCS + rTMS
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03304262/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03304262/ICF_001.pdf